CLINICAL TRIAL: NCT04824209
Title: Evaluation of Serum Markers of Pro-diabetes Inflammation in Patients With Chronic Apical Periodontitis Before and After Endodontic Treatment.
Brief Title: Serum Pro-Diabetes Inflammation Biomarkers in Patients With Apical Periodontitis.
Status: Completed | Type: Observational
Sponsor: University of Turin, Italy (Other)
Responsible Party: Sponsor
Other Study IDs: 0094485
Record Dates: First submitted 2021-03-16; First posted 2021-04-01 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Apical Periodontitis; Insulin Resistance; PreDiabetes; Diabetes; Stable
Keywords: Endodontics; Apical Periodontitis; Insulin Resistance; Diabetes; Pro-Diabetes Inflammation Markers
MeSH Terms: conditions — Periapical Periodontitis; Insulin Resistance; Prediabetic State; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples Without DNA — Blood Sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- AP group: Healthy patients between 25-55 years with Apical Periodontitis
- Control Group: Healthy patients between 25-55 years without Apical Periodontitis

SUMMARY:
Inflammation is a common factor of chronic periodontitis and diabetes. However, to date, there is no scientific evidence supporting a causal effect of the inflammation created by apical periodontitis on the onset of insulin resistance and on metabolic derangement in the condition of pre-diabetes or diabetes.

A case control study has been designed in order to evaluate serum levels of pro-diabetes inflammation factors in a sample of healthy patients between 25 and 55 years of age, with or without apical periodontitis,before endodontic treatment and at 6 and 12 months post-treatment. The aim of the study is to evaluate any relation between the presence of chronic endodontic lesions and pro-diabetes inflammation factors that can promote the onset of insulin resistance, and whether endodontic treatment can reduce these factors, thus preventing a pro-diabetes status.

DETAILED DESCRIPTION:
Healthy, consenting and informed patients of both gender under 55 years of age with apical periodontitis will be enrolled as cases. Healthy, consenting and informed patients of both gender under 55 years of age without apical periodontitis will be enrolled as control subjects. The study has been designed to assess the serum level of TNF-α, IL-1β, IL-6, IL-8 by ELISA assay.

ELIGIBILITY:
Inclusion Criteria:

* 25-55 years, healthy

Exclusion Criteria:

* under 25 years, over 55 years, patients with systemic or oral diseases or patients who underwent other dental treatments in the previous 6 months

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Dental Hospital
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2021-02-09 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2023-04-25 (Actual)

PRIMARY OUTCOMES:
Variation in pro-diabetes inflammation markers over time upon endodontic intervention. | Baseline serum levels of selected pro-diabetes inflammation markers in control group and AP group.
  Dosage of TNF-α, IL-1β, IL-6, IL-8 (pg/mL) in serum(ng/10^6 platelets) by ELISA assay.
Variation in pro-diabetes inflammation markers over time upon endodontic intervention. | Serum levels of selected pro-diabetes inflammation markers at 6 months after endodontic treatment and in control group.
  Dosage of TNF-α, IL-1β, IL-6, IL-8 (pg/mL) in serum by ELISA assay.
Variation in pro-diabetes inflammation markers over time upon endodontic intervention. | Serum levels of selected pro-diabetes inflammation markers at 12 months after endodontic treatment and in control group.
  Dosage of TNF-α, IL-1β, IL-6, IL-8 (pg/mL) in serum by ELISA assay.

CONTACTS AND LOCATIONS:
Overall Officials: Damiano Pasqualini, DDS Ass Pro, Principal Investigator — Endodontics, Department of Surgical Sciences - Univeristy of Turin
Locations (2):
- Italy (2):
  - Department of Oncology - University of Turin, Turin
  - Endodontics, Department of Surgical Sciences - Univeristy of Turin, Turin